CLINICAL TRIAL: NCT03833505
Title: Evaluation of Relationship Between Enterobius Vermicularis Infection and Bruxism in Children
Brief Title: Enterobius Vermicularis and Bruxism in Children
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Kadriye Görkem Ulu Güzel, Assistant Prof, Aydin Adnan Menderes University
Other Study IDs: 2017/003-24.03.2017
Record Dates: First submitted 2019-01-05; First posted 2019-02-07 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Bruxism, Sleep
MeSH Terms: conditions — Sleep Bruxism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1,: E. vermicularis-positive
  Interventions: Other: Bitestrip
- Group 2: E. vermicularis-negative
  Interventions: Other: Bitestrip

INTERVENTIONS:
Other: Bitestrip — The parents of the patients were asked to complete a survey that included questions about the demographic data, medical history of the patient, clinical findings of E. For diagnosis of sleep bruxism, a single-use BiteStrip® device (Up2dent, Inc.), including an electromyographic electrode, small display screen and lithium cell, was used to record the increased electromyographic activity of the masticatory muscles during sleep and bruxism, other harmful oral habits, family life and habits.

SUMMARY:
Background. Bruxism is an involuntary, non-functional activity of the masticatory system, and is frequently seen in childhood. Bruxism has many aetiologies, like malocclusion, psychological factors, allergies and gastrointestinal disorders.

Aim. To investigate the relationship between Enterobius vermicularis infection and bruxism in children.

DETAILED DESCRIPTION:
Bruxism has many aetiologies, like occlusal interferences, malocclusion, malnutrition, psychological factors, allergies and gastrointestinal disorders. Among these gastrointestinal disorders, are various intestinal parasitic infections.

Given the controversy surrounding the potential association between bruxism and intestinal parasitic infestations, both important health issues, this study sought to evaluate the relationship between E. vermicularis infection and bruxism in E. vermicularis-positive and E. vermicularis-negative 3-10-year-olds children with bruxism.

ELIGIBILITY:
Inclusion Criteria:

* Teeth-grinding at least once a week in the last 3 months before recruitment according to the criteria established by the American Academy of Sleep Medicine (AASM)
* Angle class I occlusion
* Mesial step occlusion according to flush terminal plane.

Exclusion Criteria:

* Treated with anti-helminthic drugs in the last 2 months before recruitment
* Drugs used that could affect the central nervous system and prevent sleep (sedatives, anti-depressants, neuroleptics, anti-muscarinics, selective serotonin re-uptake inhibitors)
* Sleep disorders (snoring, insomnia, obstructive sleep apnoea, restless leg syndrome, sleep-related epilepsy)
* Psychiatric or neurological disorders
* Upper respiratory system obstruction (last 15 days),
* Any systemic disease;
* Teeth erosion due to internal (reflux) or external (acidic drinks) factors
* Dermatological problems, associated with the use of BiteStrip (Up2dent, Inc., Pulheim, Germany);
* Unsuitable skin structure;
* Previously diagnosed and treated for bruxism;
* Angle class II or class III occlusion

Ages: 3 Years to 10 Years | Sex: All
Age Groups: Child
Study Population: The study included E. vermicularis-positive (Group 1, n =13) and E. vermicularis-negative (Group 2: n = 13) children aged between 3-10 years, who were admitted to Aydın Adnan Menderes University Faculty of Medicine Paediatric Gastroenterology Clinic.
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2018-05-20 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
Survey | 24.03.2017-20.05.2018
  The parents of the patients were asked to complete a survey that included questions about the demographic data, medical history of the patient, clinical findings of E. vermicularis and bruxism, other harmful oral habits, family life and habits.

SECONDARY OUTCOMES:
Oral examination | 24.03.2017-20.05.2018
  The patients who had a teeth-grinding habit were invited to, our clinic for clinical evaluation of bruxism. Patients were examined under a reflector light with inspection, palpation and mirror-sond. The extraoral examination evaluated mandibular asymmetry, joint sounds, deviation/deflection during opening/closing actions, sensitivity to palpation of masticatory muscles and pain/tenderness, sensitivity to palpation of the temporomandibular joint and masseter muscle hypertrophy10. The intraoral examination assessed the presence of wear facets on the teeth, according to a modification of the method by Johansson. The assessed teeth included primary incisors, canines and molars, permanent incisors and lower first molars. Scores were calculated as follows: 0 = no wear (none); 1 = enamel wear only (mild); 2 = enamel and dentin wear (moderate); 3 = significant loss of tooth structure (severe).

OTHER OUTCOMES:
BiteStrip | 24.03.2017-20.05.2018
  For diagnosis of sleep bruxism, a single-use BiteStrip® device (Up2dent, Inc.), including an electromyographic electrode, small display screen and lithium cell, was used to record the increased electromyographic activity of the masticatory muscles during sleep.

CONTACTS AND LOCATIONS:
Overall Officials: K. Görkem Ulu Güzel, Study Director — ADU Faculty of Dentistry Paediatric Dentistry Department
Locations (1):
- Adnan Menderes University, Faculty of Dentistry, Department of Pediatric Dentistry, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diaz-Serrano KV, da Silva CB, de Albuquerque S, Pereira Saraiva Mda C, Nelson-Filho P. Is there an association between bruxism and intestinal parasitic infestation in children? J Dent Child (Chic). 2008 Sep-Dec;75(3):276-9. PMID 19040814
- [Background] Mistry P, Moles DR, O'Neill J, Noar J. The occlusal effects of digit sucking habits amongst school children in Northamptonshire (UK). J Orthod. 2010 Jun;37(2):87-92. doi: 10.1179/14653121042939. PMID 20567031
- [Background] Tehrani MH, Pestechian N, Yousefi H, Sekhavati H, Attarzadeh H. The Correlation between Intestinal Parasitic Infections and Bruxism among 3-6 Year-Old Children in Isfahan. Dent Res J (Isfahan). 2010 Summer;7(2):51-5. PMID 22013457
- [Background] Bortoletto CC, Cordeiro da Silva F, Salgueiro Mda C, Motta LJ, Curiki LM, Mesquita-Ferarri RA, Fernandes KP, Bussadori SK. Evaluation of electromyographic signals in children with bruxism before and after therapy with Melissa Officinalis L-a randomized controlled clinical trial. J Phys Ther Sci. 2016 Mar;28(3):738-42. doi: 10.1589/jpts.28.738. Epub 2016 Mar 31. PMID 27134350
- [Background] Shochat T, Gavish A, Arons E, Hadas N, Molotsky A, Lavie P, Oksenberg A. Validation of the BiteStrip screener for sleep bruxism. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2007 Sep;104(3):e32-9. doi: 10.1016/j.tripleo.2007.03.009. Epub 2007 Jul 6. PMID 17618147
- [Background] Emodi-Perlman A, Eli I, Friedman-Rubin P, Goldsmith C, Reiter S, Winocur E. Bruxism, oral parafunctions, anamnestic and clinical findings of temporomandibular disorders in children. J Oral Rehabil. 2012 Feb;39(2):126-35. doi: 10.1111/j.1365-2842.2011.02254.x. Epub 2011 Sep 15. PMID 21916926
- [Background] Johansson A, Haraldson T, Omar R, Kiliaridis S, Carlsson GE. A system for assessing the severity and progression of occlusal tooth wear. J Oral Rehabil. 1993 Mar;20(2):125-31. doi: 10.1111/j.1365-2842.1993.tb01596.x. PMID 8468624
- [Background] Karakis D, Dogan A. The craniofacial morphology and maximum bite force in sleep bruxism patients with signs and symptoms of temporomandibular disorders. Cranio. 2015 Jan;33(1):32-7. doi: 10.1179/2151090314Y.0000000009. Epub 2014 Jun 3. PMID 25547142
- [Background] Van Wyk JA, Van Rensburg LJ, Heitmann LP. Schistosoma mattheei infection in cattle: the course of the intestinal syndrome, and an estimate of the lethal dose of cercariae. Onderstepoort J Vet Res. 1997 Mar;64(1):65-75. PMID 9204506
- [Result] Karakis D, Dogan A, Bek B. Evaluation of the effect of two different occlusal splints on maximum occlusal force in patients with sleep bruxism: a pilot study. J Adv Prosthodont. 2014 Apr;6(2):103-8. doi: 10.4047/jap.2014.6.2.103. Epub 2014 Apr 22. PMID 24843394